CLINICAL TRIAL: NCT05261828
Title: Efficacy of a Short Multidisciplinary Education and Rehabilitation Program for Patients With Subacute and Chronic Low Back Pain (LBP)
Acronym: LOMBAFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP200142; 2020-A02601-38 (Other: ID-RCB Number)
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Non Specific Low Back Pain
Keywords: low back pain; activity limitations; disability; rehabilitation; physiotherapy; exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Educational Status; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Short multidisciplinary program including education and rehabilitation and a personalized follow-up program
  Interventions: Behavioral: Education and rehabilitation associated with personalized follow-up
- B (Active Comparator): Reassuring messages and advices in agreement with the current recommendations.
  Interventions: Behavioral: Reassuring messages and advices

INTERVENTIONS:
Behavioral: Education and rehabilitation associated with personalized follow-up — short multidisciplinary program including education and rehabilitation and a personalized follow-up for patients with subacute and chronic low back pain
  Arms: A
Behavioral: Reassuring messages and advices — Reassuring messages and advices in agreement with current recommendations
  Arms: B

SUMMARY:
The main purpose of this study is to assess the clinical efficiency of an intervention including a short multidisciplinary program of education and rehabilitation and a personalized follow-up, in patients with subacute and chronic low back pain and no severe disability. The secondary objectives are:

* to assess the capacity of the program to modify and reduce the risk factors for evolution of patients towards a severe disability,
* to estimate the cost-utility ratio of the intervention.

DETAILED DESCRIPTION:
Non-specific low back pain (LBP) is the leading cause of years lived with disability worldwide. Subacute LBP is commonly defined as back pain lasting between 6 weeks and 3 months, chronic LBP as pain that persists for 3 or more months. In its most severe forms, subacute and chronic LBP can lead to severe disability that combines physical and psychological deconditioning, limitations in basic and complex activities of daily living, professional exclusion and social marginalization.

The direct and indirect medical and economic cost of chronic LBP is major for society.

Since the eighties, the bio-psycho-social approach has emerged for the treatment of people with chronic LBP and has led to multidisciplinary functional restoration (FR) programs that include physical activity, exercises, education, occupational therapy and psychological and social rehabilitation. However, the efficiency of these programs is inconsistent and their cost-effectiveness is criticized.

As FR programs are by definition standardized, the treatment of chronic LBP remains poorly stratified. However, interest in stratified therapeutic strategies has recently emerged and shown promising results. To date, in France, only semi-intensive (<100h) or intensive (>100h) FR programs dedicated to severely disabled patients with chronic LBP have been assessed The investigators' main hypothesis is that an intervention consisting in a short multidisciplinary program including education and rehabilitation and a personalized follow-up could reduce the activity limitations of not severely disabled patients with subacute and chronic LBP.

The investigators' secondary hypothesis is that such an intervention could also reduce the main risk factors for evolution of patients with LBP towards a severe disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subacute or chronic nonspecific low back pain (current episode duration ≥ 6 weeks), resistant to outpatient management, and including patients with radiculopathy as long as low back pain is predominant over pain in the lower extremity.
* Patients with less than 30 days off work (declarative) for low back pain in the previous year and involved in a professional activity at the time of inclusion.
* Patients manifesting fears and false beliefs and/or dramatization: to be included, the patient will have to answer yes to one of the following two questions:

  * Are you afraid to move?
  * Are you afraid you will never get out of it?
* Patients eligible for a rehabilitation exercise program
* informed and written consent to participate

Exclusion Criteria

* Age < 18 years,
* Insufficient French language proficiency.
* Patients having followed a multidisciplinary rehabilitation program for their low back pain in the 3 months preceding inclusion.
* Patients who have had lumbar spine surgery within the last 12 months.
* Pregnancy in progress.
* No affiliation with a health insurance program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
low back pain activity limitation | 3 months
  Variation in the level of low back pain- activity limitation assessed by the Roland-Morris self-administered questionnaire (0, no limitation and 24, maximum limitation)

SECONDARY OUTCOMES:
low back pain activity limitation | 6 and 12 months.
  Variation in the level of low back pain activity limitation assessed by the Roland-Morris self-administered questionnaire (0, no limitation and 24, maximum limitation)
fears and beliefs about work | 3 months
  Variation in the level of fears and beliefs about work assessed by the work sub score of the self-administered Fear-Avoidance Beliefs Questionnaire (FABQ) (0, no fears and beliefs and 24, maximum fears and beliefs)
fears and beliefs about physical activity | 3 months
  Variation in the level of fears and beliefs about physical activity assessed by the physical activity sub score of the self-administered Fear-Avoidance Beliefs Questionnaire (FABQ) (FABQ), (0, no fears and beliefs and 42, maximum fears and beliefs)
days off work | 3 and 12 months
  Number of "days off work" reported by the patient
low back pain | 3 months
  Variation in the mean intensity of low back pain over the last 48 hours assessed on a self-administered numerical scale (0, no pain and 100,maximum pain)
radicular pain | 3 months
  Change in mean intensity of radicular pain over the last 48 hours assessed on a self-administered numerical scale (0, no pain and 100,maximum pain)
cost-utility ratio | 12 months
  Incremental cost-utility ratio

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra ROREN, PhD, Principal Investigator — APHP
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No